CLINICAL TRIAL: NCT00528944
Title: Single-Breath Measurement Underestimates Ventilatory Volume According to Emphysema Severity
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAB6328
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Emphysema
Keywords: alveolar volume; pulmonary function testing; emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort A: Patients with obstructive defects and radiological evidence of emphysema
- Cohort B: Patients with obstructive ventilatory defects and no radiological evidence of emphysema
- Cohort C: Non-smokers without obstructive ventilatory defects or history of cardiopulmonary disease

SUMMARY:
Although single breath helium (He) dilution measurement (VASB) is currently used in pulmonary function laboratories to assess functional alveolar volume and diffusing capacity for carbon monoxide, the extent to which VASB reflects ventilatory and thoracic volume has not been prospectively determined in emphysema. We hypothesized that VASB underestimates rebreathe helium dilution volume (VARB), and plethysmographic volume (VApleth) as clinical and physiologic severity of emphysema increases.

DETAILED DESCRIPTION:
VASB, VARB, and VApleth were measured in 52 consecutive stable outpatients with clinical and radiographic emphysema. Thirteen patients with an obstructive ventilatory defect without emphysema (OVD) and 18 normal controls were similarly studied. All subjects underwent spirometry followed by whole body plethysmography and He dilution volume measurements; VASB and VARB order was randomized.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients between the ages of 18 and 81 years referred to the Columbia University Medical Center Pulmonary Diagnostic Unit between 1/18/06 and 7/30/07 for full pulmonary function evaluation, and with an obstructive ventilatory defect on spirometry, were considered eligible.

Exclusion Criteria:

* Patients who did not want to undergo the re-breathe diffusing capacity testing
* Patients who could not give informed consent;and
* Patients who were too physically compromised to undergo full testing including the re-breathe maneuver as deemed by our technicians.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective trial in all outpatients with emphysema referred for full pulmonary function testing to the pulmonary diagnostic unit.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Difference between DLCO SB alveolar volume and the total lung volume measurement from plethysmography | 10 seconds
  To test the hypothesis that DLCO SB underestimates DLCO derived by the re-breathe DLCO maneuver, and that VA SB similarly underestimates VA RB. Alveolar volume derived with the two maneuvers will be compared with body plethysmography, the gold standard of total lung volume measurement in patients with emphysema.
Difference between DLCO RB alveolar volume and the total lung volume measurement from plethysmography | 10 seconds
  To test the hypothesis that DLCO SB underestimates DLCO derived by the re-breathe DLCO maneuver, and that VA SB similarly underestimates VA RB. Alveolar volume derived with the two maneuvers will be compared with body plethysmography, the gold standard of total lung volume measurement in patients with emphysema.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Basner, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Cardiopulmonary, Sleep and Ventilatory Disorders Center, New York, New York, United States